CLINICAL TRIAL: NCT07114497
Title: Investigation of miRNA Expression Profiles in Human Degenerated Intervertebral Disc Tissues
Acronym: MIRADISC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Collaborators: Canakkale 18 Mart University Health Research and Application Hospital (Unknown)
Responsible Party: Principal Investigator, DAMLA AYKORA, Principal Investigator, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: TSA-2025-5076; TSA-2025-5076 (Other Grant/Funding Number: Çanakkale Onsekiz Mart University Experimental Research Coordination Unit)
Record Dates: First submitted 2025-07-31; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Degeneration Disc Intervertebral; miRNA
Keywords: Disc degeneration; miRNA
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Degenerated Disc Group (IVDD Group) (Experimental): This group consists of patients diagnosed with lumbar disc herniation (LDH) who are scheduled for lumbar microdiscectomy (LMD) surgery due to intervertebral disc degeneration (IVDD).
  Interventions: Diagnostic Test: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines; Diagnostic Test: excised; Diagnostic Test: Diagnostic work up
- Non-degenerated Disc Control Group (Experimental): This group includes patients undergoing spinal surgery (decompression or fusion) due to vertebral fractures, with no signs of intervertebral disc degeneration. Only patients without degenerative changes on imaging will be included.
  Interventions: Diagnostic Test: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines; Diagnostic Test: excised; Diagnostic Test: Diagnostic work up

INTERVENTIONS:
Diagnostic Test: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines — During surgery, degenerated intervertebral disc tissues will be collected under sterile conditions and stored at -80°C in cryotubes. miRNA expression profiles will be analyzed using rt-PCR. Candidate miRNAs are selected based on databases such as miRBase, miRTar, and miRDB.
Diagnostic Test: excised — Intervertebral disc tissues that are not degenerated will be collected during surgery and stored in the same manner as in the IVDD group. These samples will be used for comparative analysis of miRNA expression via rt-PCR to serve as the control baseline.
Diagnostic Test: Diagnostic work up — During surgery, degenerated intervertebral disc tissues will be collected under sterile conditions and stored at -80°C in cryotubes. miRNA expression profiles will be analyzed using rt-PCR. Candidate miRNAs are selected based on databases such as miRBase, miRTar, and miRDB.

SUMMARY:
Aim of the Study:

The aim of this study is to determine the expression levels of candidate microRNAs (miRNAs) expressed in human degenerated intervertebral disc tissues. In line with this objective, our specific goals are outlined below:

Objectives:

Objective 1:

To include patients diagnosed with lumbar disc herniation (LDH) who are scheduled for lumbar microdiscectomy (LMD), and patients diagnosed with vertebral fractures who are scheduled for decompression or fusion surgeries, by obtaining informed consent in accordance with ethical standards.

Objective 2:

To collect degenerated intervertebral disc tissues obtained during LMD or spinal cord repair surgeries into cryotubes in duplicates for real-time PCR (rt-PCR) analysis, and to store them under appropriate conditions until analysis.

Objective 3:

To identify candidate miRNAs that regulate genes associated with the pathophysiology of intervertebral disc degeneration (IVDD) using databases such as miRBase, miRTar, and miRDB.

Objective 4:

To determine the expression levels of candidate miRNAs associated with nucleus pulposus cell proliferation in human degenerated disc tissues.

Objective 5:

To determine the expression levels of candidate miRNAs associated with apoptosis of nucleus pulposus cells in human degenerated disc tissues.

Objective 6:

To determine the expression levels of candidate miRNAs associated with extracellular matrix (ECM) remodeling in human degenerated disc tissues.

Objective 7:

To determine the expression levels of candidate miRNAs associated with cartilaginous endplate dysfunction in human degenerated disc tissues.

Objective 8:

To determine the expression levels of candidate miRNAs associated with annulus fibrosus degeneration in human degenerated disc tissues.

Objective 9:

To determine the expression levels of candidate miRNAs associated with inflammatory processes in human degenerated disc tissues.

Objective 10:

To compare the expression levels of each candidate miRNA identified in degenerated disc tissues with those found in non-degenerated disc tissues obtained during spinal cord repair surgeries.

ELIGIBILITY:
Inclusion Criteria:

* ıvdd surgery, fracture suregery

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-10-12 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
disc degeneration | 1 year
  degeneration level assessment

SECONDARY OUTCOMES:
disc degeneration | 1 year
  degeneration level assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz Mart University, Çanakkale, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided